CLINICAL TRIAL: NCT04632238
Title: Coaching Performance Driven Practice Change in the Context of Value Based Purchasing Under New York Medicaid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); New York State Office of Addiction Services and Supports (Unknown); UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-00776
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Opioid-use Disorder; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Trial (SW-RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Metrics-driven quality improvement (MDQI) intervention (Experimental)
  Interventions: Behavioral: Metrics-driven quality improvement (MDQI)

INTERVENTIONS:
Behavioral: Metrics-driven quality improvement (MDQI) — The intervention broadly consists of training and coaching to clinic staff and leadership on 1) clinical quality measure monitoring; 2) clinical practice process change management; and 3) use of tools for shared decision making and patient treatment progress monitoring.
  Arms: Metrics-driven quality improvement (MDQI) intervention

SUMMARY:
This project will develop and test quality measures for and a facilitation model to help addictions treatment clinics increase use of medicines for opioid use disorders, retain clients longer in care, and help more people move into successful recovery. At the end of the project, we will have developed specific training and coaching protocols as well as electronic clinical support tools to guide quality improvement that can be disseminated within New York and the rest of the country.

The study will test a clinic-level intervention that uses external facilitators to provide guidance to addictions clinics and contain three key components: 1) training on data driven management; 2) training and guidance on patient-centered care and OUD medication; and 3) electronic tools for shared decision making and patient progress monitoring.

DETAILED DESCRIPTION:
There will be 4 sources of data examined in this study: 3 at the patient level and 1 at the staff level. The sources of patient data include: 1) State administrative data from all clients receiving treatment at the enrolled clinics (~7,950); 2) a subsample (1,200) who will be recruited directly from the clinics to complete patient-reported outcome assessments, and 3) treatment progress data for clients will also be collected.

For our administrative source of data, a final study population of approximately 7,950 individuals who are receiving treatment in the 30 enrolled outpatient treatment clinics for OUD is anticipated. Clinics will be located in the New York City metropolitan region (including Nassau, Westchester, and Rockland counties) and the Capital Region (including Albany, Rensselaer, Saratoga, Montgomery, Schenectady, and Schoharie counties). Staff at each enrolled clinic will also be interviewed and surveyed.

ELIGIBILITY:
Inclusion Criteria:

* Substance use disorder clinics in the regions surrounding New York City and the New York Capital Region with annual census of 50 or greater.
* All staff and patients from participating clinics will be eligible to participate in the study.
* Inclusion in the analyses using administrative data will be limited to those enrolled in Medicaid and not co-insured with Medicare (individuals ages greater than 64 and those with Federally determined disability).

Exclusion Criteria:

* Patients who are not working/being treated at substance use disorder clinics with less than 50 clients per year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7950 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in clinic-level rates of initiation to OUD medications | Assessed from commencement of the trial in Year 1 of the study to the conclusion of the trial in Year 4 of the study.
Change in clinic-level rates of adherence to OUD medications | Assessed from commencement of the trial in Year 1 of the study to the conclusion of the trial in Year 4 of the study.
Retention in Care | Assessed from commencement of the trial in Year 1 of the study to the conclusion of the trial in Year 4 of the study.
  Clinic rates of 6-month client retention in care
Change in Incidence of Overdoses | Assessed from commencement of the trial in Year 1 of the study to the conclusion of the trial in Year 4 of the study.
Change in Incidence of Substance Use-Related Hepatitis C Infection | Assessed from commencement of the trial in Year 1 of the study to the conclusion of the trial in Year 4 of the study.
Change in Number of Emergency Room Visits | Assessed from commencement of the trial in Year 1 of the study to the conclusion of the trial in Year 4 of the study.
Change in Health Status | Assessed from the start of each clinic in the intervention to 1 year post-intervention
  Change in health status is measured by the first item of the SF-12 Health Survey: "In general, would you say your health is: 1 - excellent, 2 - very good, 3 - good, 4 - fair, 5 - poor". Scores range from 1-5, with a higher score indicating worse health.

SECONDARY OUTCOMES:
Cost of treatment | Assessed from commencement of the intervention at each clinic to 1 year post-intervention
  Cost of the intervention to the clinic
Change in clinic-level rates of clients with Severe OUD | Assessed from commencement of the intervention at each clinic to 1 year post-intervention
  As indicated by daily use and/or injection drug use as indicated in state administrative admission data
Change in clinic level-rates of clients identified as homeless | Assessed from commencement of the intervention at each clinic to 1 year post-intervention
  As indicated in state administrative admission data
Change in clinic-rates of clients with co-existing psychiatric disorder as indicated in state administrative admission data | Assessed from commencement of the intervention at each clinic to 1 year post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charles Neighbors, PhD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - Samaritan Rockland - Outpatient Program, Blauvelt, New York
  - Samaritan Queens - Jamaica IOP, Jamaica, New York
  - Samaritan Daytop Village Harlem - Outpatient Program, New York, New York
  - Upper Manhattan Addiction Treatment Services Program, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article resulting from surveys only, after deidentification (text, tables, figures, and appendices), will be available. Client outcome data from State administrative data files will not be available for sharing due to the nature of the data security agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Charles.Neighbors@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] O'Grady MA, Lincourt P, Greenfield B, Manseau MW, Hussain S, Genece KG, Neighbors CJ. A facilitation model for implementing quality improvement practices to enhance outpatient substance use disorder treatment outcomes: a stepped-wedge randomized controlled trial study protocol. Implement Sci. 2021 Jan 7;16(1):5. doi: 10.1186/s13012-020-01076-x. PMID 33413493